CLINICAL TRIAL: NCT03628196
Title: Assessing the Feasibility and Effectiveness of a Nutrition-Focused Quality Improvement Program (QIP) in Outpatient Clinics Affiliated With an Academic Health System
Brief Title: A Nutrition-Focused QIP in Outpatient Clinics
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: HA35
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Quality Improvement Program Basic and Enhanced Phase: Patients that meet the eligibility criteria and participate in the QIP.
- Retrospective Group: Patients seen a year prior to the QIP period at the clinic but that did not participate in the QIP.
- Concurrent Group: Patients seen during the QIP period at the clinic but that did not participate in the QIP.

SUMMARY:
A nutrition-focused QIP will be implemented with a primary assessment of QIP feasibility, patient health and economic outcomes as well as patient and provider experience data. A 2-phased QIP study group will be prospectively enrolled from outpatient clinics affiliated with the USC health system and compared with historical and concurrent control groups.

ELIGIBILITY:
QIP Group

Inclusion Criteria:

* Poor nutritional status
* 2 or more chronic conditions (other than those listed as exclusions)
* Estimated life expectancy of 90 days or greater
* Able to consume foods and beverages orally
* Literate and willing to sign informed consent form

Exclusion Criteria:

* Pregnant
* Normal nutritional status
* Unable to consume foods and beverages orally
* Estimated life expectancy of less than 90 days
* Severe dementia or delirium and no dedicated caregiver to assure compliance with QIP study requirements
* Uncontrolled eating disorder, significant neurological or psychiatric disorder (including substance abuse), or other conditions that may interfere with study product consumption or compliance
* Known allergy or intolerance to any ingredient found in ONS products recommended in QIP

Retrospective and Concurrent groups eligibility are reflective of the QIP eligibility criteria however, the timeframe differs.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in participating outpatient centers of the USC health system.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Health Resource Utilization | Enrollment to 90 days
  Number of visits

SECONDARY OUTCOMES:
Change in Medication Usage | Enrollment to 90 days
  Obtained from EMR
Quality of Life (QOL) SF-12 | Enrollment to 90 days
  Patient reported (QOL) questionnaire
Satisfaction with Nutritional Care including screening, education and oral nutrition supplementation recommendations and follow up. | Enrollment to 90 days
  QIP patient completed 5-point Likert scale
Nutrition Care Program Health Care Professionals (HCPs) Survey | 90 days
  11, 5-point Likert scale questions, scaled in the positive direction; 9 program description questions

CONTACTS AND LOCATIONS:
Overall Officials: Suela Sulo, PhD, Msc., Study Chair — Abbott Nutrition; Kurt Hong, MD, PhD, FACN, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Keck Medical Center of USC, Internal Medicine and Family Medicine Clinics, Los Angeles, California
  - Pasadena - USC Healthcare Center, Pasadena, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hong K, Sulo S, Wang W, Kim S, Huettner L, Taroyan R, Kerr KW, Kaloostian C. Nutrition Care for Poorly Nourished Outpatients Reduces Resource Use and Lowers Costs. J Prim Care Community Health. 2021 Jan-Dec;12:21501327211017014. doi: 10.1177/21501327211017014. PMID 34009072